CLINICAL TRIAL: NCT06019832
Title: Analysis of Varus Collapse in Obese Patients With Stem and Non-Stem Tibial Components Following Primary Total Knee Arthroplasty
Acronym: SvNS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jacob M. Elkins (Other)
Responsible Party: Sponsor-Investigator, Jacob M. Elkins, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202303366
Record Dates: First submitted 2023-08-24; First posted 2023-08-31 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Aseptic Loosening; Varus Collapse
MeSH Terms: conditions — Obesity | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A: Stemmed Tibial Implant (Active Comparator): This study group will receive a stemmed tibial implant as part of their TKA.
  Interventions: Procedure: Total Knee Arthroplasty (TKA); Device: Stemmed Tibial Implant
- Group B: Non-Stemmed Tibial implant (Active Comparator): This study group will receive a non-stemmed tibial implant as part of their TKA.
  Interventions: Procedure: Total Knee Arthroplasty (TKA); Device: Non-stemmed tibial implant

INTERVENTIONS:
Procedure: Total Knee Arthroplasty (TKA) — Both study arms will undergo TKA
Device: Stemmed Tibial Implant — A stemmed tibial implant.
  Arms: Group A: Stemmed Tibial Implant
Device: Non-stemmed tibial implant — A non-stemmed tibial implant.
  Arms: Group B: Non-Stemmed Tibial implant

SUMMARY:
The purpose of this study is to compare rates of varus collapse, aseptic loosening, and implant failure in female obese patients undergoing total knee arthroplasty (TKA) and will review the degree of influence of stemmed tibial components versus non-stemmed tibial components on varus collapse and aseptic loosening, a consequence of implant micromotion.

DETAILED DESCRIPTION:
The purpose of this study is to identify varus collapse, aseptic loosening, and implant failure in female obese patients undergoing total knee arthroplasty (TKA). In addition, this study will review the degree of influence of stemmed tibial components versus non-stemmed tibial components on varus collapse and aseptic loosening, a consequence of implant micromotion.

Female patients age 40 and older with BMI of 35 kg/m2 and above will be randomized into two groups: the non-stem tibial component (control group) and the stem tibial component (treatment group). Previous studies done in the past in normal weight patients showed that there is little or no advantage in using the stem tibial implants over the non-stem ones. Theoretically, biomechanical studies have suggested that there may be improved fixation and load distribution with the use of stem tibial implants. Thus, it is necessary to see if there is any difference between both implant options among female patients who have the highest incidence of varus collapse. In terms of design, the stem tibial implants are slightly longer than the non-stem ones. They are designed to extends deeper into the tibia to enhance fixation and improve load distribution. The use of either stem tibial implants is usually based on patients' characteristics and surgeons' preference.

Following informed consent, standard perioperative patient-reported metrics will be collected (Knee Injury and Osteoarthritis Outcome Score for Joint Replacement [KOOS-JR], American Knee Society score, and Patient-Reported Outcome Measurement Information System 10 [PROMIS-10]) before surgery and after surgery (3-6 weeks, 8-12 weeks, 1 year, 3 years, and 5 years). After surgery, study participants will receive routine surgical care which includes two knee radiographs at 8-12 weeks and one year. In addition to this, the study participants will be evaluated at 3 years, and 5 years postoperative periods where they will complete routine PROMs as listed above and have knee radiographs during each visit.

ELIGIBILITY:
Inclusion criteria:

* Female adult patients with severe osteoarthritis scheduled to have primary total knee arthroplasty
* Age 40 or older
* 35 kg/m2 and above
* Only patients from the PI's clinic will be included.
* Women who are still menstruating and are currently on contraceptives and women who are in menopause.

Exclusion Criteria:

* Patients who have some active local or widespread infection (including secondary or inflammatory osteoarthritis)
* medical conditions that put them at risk of complications or death during and after the study would not be eligible for surgery
* Patients with previous knee surgery on arthroplasty site will be excluded
* Pregnant patients and women who are capable of getting pregnant

Ages: 40 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Varus Collapse | up to 5 years post surgery
  The investigators will track rate of varus collapse.
Aseptic loosening | up to 5 years post surgery
  The investigators will track rates of aseptic loosening.

CONTACTS AND LOCATIONS:
Locations (1):
- Iowa Health Care Medical Center North Liberty, North Liberty, Iowa, United States